CLINICAL TRIAL: NCT06328049
Title: A Prospective, Single-arm, Exploratory Clinical Study of Trilaciclib Combined With Chemotherapy in the Treatment of Advanced Non-small Cell Lung Cancer
Brief Title: A Study of Trilaciclib Combined With Chemotherapy in the Treatment of NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Taixing People's Hospital (Other)
Responsible Party: Principal Investigator, Liu Yangchen, Director, Taixing People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HSKY-033
Record Dates: First submitted 2024-03-13; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: NSCLC
MeSH Terms: interventions — trilaciclib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trilaciclib plus chemotherapy (Experimental): Patients with lung adenocarcinoma were treated with Trilaciclib (240mg/m2, d1, within 4 hours before each chemotherapy) combined with pemetrexed and carboplatin (dose according to the guideline recommendation, d1, Q3W). "For squamous lung cancer, Trilaciclib (d1, 240mg/m2, 4 hours before each chemotherapy) plus paclitaxel/albumin-bound paclitaxel plus carboplatin (dose according to guideline recommendation, d1), Q3W." In the second cycle, patients were left to their own discretion with or without treaclib combination therapy.
  Interventions: Drug: Trilaciclib Injection

INTERVENTIONS:
Drug: Trilaciclib Injection — Patients with lung adenocarcinoma were given Trilaciclib combined with pemetrexed and carboplatin, Q3W; For patients with lung squamous cell carcinoma,Trilaciclib combined with paclitaxel/albumin-bound paclitaxel and carboplatin, Q3W. From cycle 2 onwards, patients chose whether to use trasylol with chemotherapy.
  Other Names: CDK4/6 inhibitors

SUMMARY:
The aim of this study is to investigate the safety and efficacy of the prophylactic use of Trilaciclib in patients with non-small cell lung cancer (NSCLC) receiving platinum-based chemotherapy, so as to provide more evidence-based medical evidence for the optimal diagnosis and treatment strategy in this population.

DETAILED DESCRIPTION:
This is a single-arm, exploratory clinical study. Eligible patients were treated with Trilaciclib before the first cycle of chemotherapy, and their peripheral blood samples were tested on days 3,7,14,21±1 after chemotherapy. At the same time, the incidence of FN, the use of antibiotics, the safety, the number of patients who delayed the second cycle of treatment, the number of patients who reduced the dose of chemotherapy, the number of patients who reduced the dose of chemotherapy due to neutropenia, and the number of patients who discontinued chemotherapy were observed.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years old (including 18 years old)，regardless of gender；
* ECOG-PS score of 0-1,；
* expected survival≥12 weeks；
* There was no tumor deterioration in the 2 weeks prior to study drug treatment.
* Advanced non-small cell lung cancer without systemic chemotherapy.
* At least one tumor lesion with a maximum diameter ≥10 mm (short diameter ≥15 mm if it is a lymph node) that could be measured accurately at baseline according to RECIST1.1 criteria. Baseline tumor imaging was performed within 28 days before the first dose.
* Women of childbearing age should use appropriate contraception and should not breastfeed from screening until 3 months after discontinuation of study treatment.
* Male subjects should use barrier contraception (i.e., condoms) for 3 months from screening until discontinuation of study treatment.
* All subjects voluntarily participated and signed the informed consent form in person.

Exclusion Criteria:

* Uncontrolled ischemic heart disease or clinically significant congestive heart failure (NYHA class III or IV);
* stroke or cardio-cerebrovascular event within 6 months before enrollment;
* QTcF interval > 480msec at screening or > 500msec for patients with implanted ventricular pacemakers;
* Previous hematopoietic stem cell or bone marrow transplantation;
* Allergy to the study drug or its components;
* Others considered by the investigator to be unsuitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-02-10 (Estimated); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of febrile neutropenia (FN) | during Trilaciclib plus chemotherapy assessed up to 21 days
  Incidence of febrile neutropenia in the first treatment cycle

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Up to 2 years
  Occurrence and severity of AEs by NCI CTCAE v5.0
Antibiotic Use rate | during Trilaciclib plus chemotherapy assessed up to 21 days
  Antibiotic Use rate in the first treatment cycle
Number of medication delays | At the end of Cycle 1 (each cycle is 28 days)
  Number of delays in the second treatment cycle due to myelosuppression
Number of chemotherapy dose reductions | At the end of Cycle 1 (each cycle is 28 days)
  Number of chemotherapy dose reductions in the second treatment cycle due to myelosuppression

CONTACTS AND LOCATIONS:
Overall Officials: liu C yang, M.D., Principal Investigator — Taixing People's Hospital
Locations (1):
- Taixing People's Hospital, Taishing, Jiangsu, China